CLINICAL TRIAL: NCT04169750
Title: Home-based EXergames To impRove cognitivE Function in MUltiple Sclerosis: the EXTREMUS Study. A Multicenter, Randomized, Single-blind Non-inferiority Trial
Brief Title: Home-based EXergames To impRove cognitivE Function in MUltiple Sclerosis
Acronym: EXTREMUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Camillo Hospital, Rome (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); Fondazione Italiana Sclerosi Multipla (Other); Rehabilitation Unit 'Mons. L. Novarese' Hospital, Moncrivello (VC), IT (Unknown); University of Chieti (Other)
Responsible Party: Principal Investigator, Luca Prosperini, Principal Investigator, San Camillo Hospital, Rome
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/R/22
Record Dates: First submitted 2019-11-03; First posted 2019-11-20 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Cognitive impairment; Exergames; Neuroplasticity; Clinical Trial
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergames (Experimental)
  Interventions: Behavioral: Exergames
- Adaptive COGNI-TRAcK (Active Comparator)
  Interventions: Behavioral: Adaptive COGNI-TRAcK
- Sham COGNI-TRAcK (Sham Comparator)
  Interventions: Behavioral: Sham COGNI-TRAcK

INTERVENTIONS:
Behavioral: Exergames — The training protocol will be delivered by the Nintendo ® Wii balance board and consists of repetitions of several games selected from the "Wii Fit Plus" package (http:// www.wiifit.com/training/balance-games.html). Each game starts at basic level, and when a certain score is reached, patients is automatically transferred to a more advanced level. Patients will be encouraged to play the next game if they have a level progress; otherwise, 10 minutes will be allocated for each game. During the first 4 weeks of training, patients will be allowed to play only "Zazen" (sitting position), "Table Tilt" and "Ski Slalom"; thereafter they will add the remaining games "Penguin Slide", "Tightrope Walk", "Balance Bubble" and "Soccer Heading".
  Arms: Exergames
Behavioral: Adaptive COGNI-TRAcK — The training protocol will be delivered by a dedicated app for mobile devices (mobile phone or tablet). The app implements three different types of exercises (each one executed for about 10 min a session), consisting in a visuo-spatial working memory task, an "operation" N-back task and a "dual" N-back task.
  The adaptive training is structured so that the exercises difficulty level will increase by one step every time the user will perform a correct exercise. On the other hand, the difficulty level will decrease by one step if the exercise is incorrect for three times in a row.
  Arms: Adaptive COGNI-TRAcK
Behavioral: Sham COGNI-TRAcK — The training protocol will be delivered by a dedicated app for mobile devices (mobile phone or tablet) as previously described for adaptive COGNI-TRAcK. However, the non-adaptive training (placebo-analogue intervention) consists in an algorithm implementing two low difficulty levels alternating every day regardless of the user's performance.
  Arms: Sham COGNI-TRAcK

SUMMARY:
Study design: Phase II, multicenter, randomized, sham-controlled, single-blind, parallel arm, multicenter study to test the hypothesis that home-based exergames is not inferior to home-based cognitive rehabilitation delivered by a software application (app) for mobile devices and both interventions are superior to a placebo-analogue cognitive intervention in improving cognitive function and reducing cognitive-motor interference in people with multiple sclerosis (MS).

Procedures: Participants will be randomized in a 1:1:1 ratio to receive an 8-week home-based training with exergames (intervention of interest) or adaptive COGNI-TRAcK (comparator intervention) or sham COGNI-TRAcK (placebo-analogue intervention). Study assessment will be done at study enrolment (baseline), at the end of the 8-week intervention period (immediate post-training, Week 8) and after 16 weeks from randomization (post-training follow-up, Week 16).

Investigational interventions:

1. Exergames: home-based repetition of several games delivered by the Nintendo © Wii Balance Board, a commercial off-the-shelf video game console for re-training of balance and postural strategies
2. Adaptive COGNI-TRAcK: adaptive (i.e. automatic adjustment of tasks difficulty) working memory training delivered by a customized application software for mobile devices to self-administer at-home
3. Sham COGNI-TRAcK: non-adaptive (i.e. constant difficulty level) working memory training delivered by the same app as afore described

Primary endpoint: changes at the Symbol Digit Modalities Test (SDMT), a measure of sustained attention and information processing speed.

Secondary endpoint: changes at the BICAMS (z-scores), a brief, practical and universal assessment tool for cognitive impairment in MS.

Additional endpoints: magnitude of cognitive-motor interference estimated as dual-task cost of balance and walking.

Sample size estimation: The investigators estimated a pre-defined 8-point non-inferiority margin, based on a significant effect of the COGNI-TRAcK in inducing an about 8-point mean increase at SDMT score (with respect to a sham intervention). Accordingly, 35 participants per arm are required to ensure, with an approximately 85%-power level, that the lower limit of a one-side 95% confidence interval will be above the pre-defined non-inferiority margin. Therefore, considering also a drop-out rate of 25%, a total of 132 subjects should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years (inclusive);
* cognitive impairment, defined as failure in the SDMT, defined as a corrected score less than 38, i.e. below the 5th percentile of normative value;
* Expanded Disability Status Scale (EDSS) score between 2.0 and 5.5;
* ability to stand upright for at least 180 seconds without any support;
* ability to understand and comply with study requirements;
* ability to provide a valid informed consent before any study procedure.

Exclusion Criteria:

* relapse in the previous 6 months;
* initiation of disease-modifying or symptomatic treatments or physiotherapy programme in the 3 months prior to study entry;
* any medication/physiotherapy changes occurring over the previous 3 months;
* significant visual impairment, defined as a Visual System scoring more than 2 at the Kurtzke Functional Systems Score;
* clinically relevant depression, defined as Beck Depression Inventory-II (BDI-II) score equal or more than 14;
* overt dementia, defined as an adjusted Mini Mental State Examination (MMSE) score equal or less than 24;
* history of epilepsy or seizures;
* any medical condition, including musculoskeletal disorders that can interfere with the study conduction.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test | Change from randomization to 8-week visit
  The participant is presented with a page headed by a key that pairs the single digits 1-9 with nine symbols. Rows below contain only symbols, the subject's task is to orally report the correct number in the spaces below. After completing the first 10 items with guidance, the subject is timed to determine how many responses can be made in 90 seconds.
  Range score: not applicable. Higher scores mean a better outcome. Explored domain: Sustained attention and information processing speed.

SECONDARY OUTCOMES:
Brief International Cognitive Assessment for Multiple Sclerosis | At randomization, 8 weeks and 16 weeks
  Brief cognitive assessment for multiple sclerosis that includes the Symbol Digit Modalities Test (SDMT) for exploring sustained attention, the initial learning trials of the second edition of the California Verbal Learning Test (CVLT2) for exploring auditory/verbal learning, and the revised Brief Visuospatial Memory Test (BVMTR) for exploring visual/spatial memory.
  Range score: not applicable. Higher scores mean a better outcome.
Stroop Color-Word Test | At randomization, 8 weeks and 16 weeks
  The test explores some aspects of executive functions and consists of naming the color of the ink of words, indicating conflicting colors as quickly as possible.
  Range score: not applicable. Higher scores mean a better outcome.

OTHER OUTCOMES:
Cognitive-Motor Interference | At randomization, 8 weeks and 16 weeks
  Dual-task cost of walking (2-Meter Walking Test) and balance (static posturography) is calculated as percentage change in scores obtained under single-task condition minus dual-task condition divided by the score under single-task condition.
  Range score: not applicable (negative values are possible). Higher scores mean a better outcome.
29-item Multiple Sclerosis Impact Scale | At randomization, 8 weeks and 16 weeks
  The Multiple Sclerosis Impact Scale (MSIS-29) is a 29-item self-administered questionnaire measuring physical and psychological impact of multiple sclerosis from the patient's perspective.
  Range score: 0 to 100. Higher scores mean worse outcome.
21-item Modified Fatigue Impact Scale | At randomization, 8 weeks and 16 weeks
  The Modified Fatigue Impact Scale (MFIS) is a 21-item self-administered questionnaire based on items derived from interviews with patients with multiple sclerosis concerning how fatigue impacts their lives; it comprises three subscales (physical, cognitive, and psychosocial functioning).
  Range score: 0 to 84. Higher scores mean worse outcome.
Work Productivity and Activity Impairment: Multiple Sclerosis | At randomization, 8 weeks and 16 weeks
  To quantify absenteeism (missing work because of health problems), presenteeism (impairment while working), overall work impairment, and daily activity impairment attributable to multiple sclerosis.
  Range score: 0 to 100. Higher scores mean worse outcome.
Time to first accidental falls | From randomization to study termination (16 weeks)
  Time to randomization to the first accidental falls reported by the participant, defined as an event which results in a person coming to rest inadvertently on the ground or floor or other lower level (WHO).
  Range score: not applicable.
Adverse events | From randomization to study termination (16 weeks)
  Any untoward medical occurrence in participants which does not necessarily have a causal relationship with the administered intervention.
  Range score: not applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Prosperini, MD, PhD, Principal Investigator — A.O. San Camillo-Forlanini
Locations (4):
- Italy (4):
  - Italian MS Foundation, Genova, GE
  - LaRiCE Lab, Don Gnocchi Foundation IRCCS, Milan, MI
  - A.O. San Camillo, MS Center, Rome, RM
  - Dept. of Rehabilitation, M.L. Novarese, Moncrivello, VC

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: After publication
Access Criteria: Upon request to PI

REFERENCES:
- [Derived] Prosperini L, Tacchino A, Ruggieri S, Brichetto G, Podda J, Anastasi D, Cardini R, Corrini C, Quartuccio ME, Alcamisi I, Di Giovanni R, Gamberini G, Grange E, Pietrolongo E, Rispoli MG, Tomassini V, Cattaneo D, Solaro C. Home-based EXergames To impRovE cognitive function in MUltiple Sclerosis (EXTREMUS). J Neurol Neurosurg Psychiatry. 2025 Oct 1:jnnp-2025-336609. doi: 10.1136/jnnp-2025-336609. Online ahead of print. PMID 41033785

DOCUMENTS (1):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04169750/Prot_000.pdf